CLINICAL TRIAL: NCT00198315
Title: A Randomized Trial Comparing Preservation of Function Status After Either Medpulser Electroporation With Intratumoral Bleomycin Therapy or Surgery in Patients With Locally Recurrent or Second Primary Squamous Cell Carcinoma of the Anterior Oral Cavity, Soft Palate, or Tonsil That Have Failed Primary Curative Therapy
Brief Title: Medpulser Electroporation With Bleomycin Study to Treat Anterior Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment was stopped based on the Data Monitoring Committee's recommendation.
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNBE-03-01; HNBE-03-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Cancer
Keywords: Squamous Cell Carcinoma; Carcinoma; Head and Neck Cancer; Oral; Soft Palate; Cancer; Medpulser; Electroporation; Local recurrent or second primary squamous cell carcinoma of anterior oral cavity, soft palate, or tonsil
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Carcinoma; Neoplasms | interventions — Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery Control (Active Comparator): Patients will receive standard of care surgical removal of their tumor.
  Interventions: Procedure: Tumor surgical excision
- MedPulser EPT with Bleomycin (Experimental): Patients who are eligible for surgical excision will receive MedPulser electroporation with injection of bleomycin sulfate into the tumor treatment area.
  Interventions: Combination Product: Medpulser electroporation with Bleomycin

INTERVENTIONS:
Combination Product: Medpulser electroporation with Bleomycin — Patients receive electroporation with injection of bleomycin sulfate at a concentration of 1 U/ml per cm3 of tumor treatment area.
  Arms: MedPulser EPT with Bleomycin
Procedure: Tumor surgical excision — Patients have their tumor surgically removed.
  Arms: Surgery Control

SUMMARY:
The purpose of the study is to evaluate Medpulser electroporation (EPT) with bleomycin with regard to local tumor recurrence, disease-free survival, and overall survival rates versus surgery in recurrent or secondary primary squamous cell carcinoma (SCC) of the anterior oral cavity, soft palate, or tonsil.

DETAILED DESCRIPTION:
Recurrent tumors in head and neck squamous cell carcinoma usually have a poor prognosis. In patients suitable for salvage surgery of their recurrent disease, the success rate for local control has been reported to be 40-50%. The surgical treatment of H&N SCC frequently results in significant loss of organ function (e.g., inability to swallow, speak, etc.) and/or permanent disfigurement. There is a compelling and unmet medical need for a local therapy that destroys tumors while preserving function status and appearance in patients with primary, recurrent, or metastatic H&N SCC.

Comparison: To compare function status at 4 months after treatment with bleomycin-EPT or surgery in patients with locally recurrent or second primary SCC of the anterior oral cavity, soft palate, or tonsil that have failed primary curative therapy and in whom surgical resection is seen as an option for disease control.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of SCC of the anterior oral cavity, soft palate or tonsil must be confirmed by histological examination of a tissue sample (e.g., biopsy) obtained within 1 month of the patient receiving the study treatment.
2. Recurrent or second primary disease in patients where surgical resection is seen as an option for disease control.
3. The length of the longest diameter of the study lesion must be < 5 cm and the calculated treatment volume must be < 60.0 cm3 (tumor volume plus a 0.5 cm margin around the tumor) for the study lesion [where treatment volume = 0.5 (A+1) (B+1)2 and where A = length of the longest diameter (cm), B = the next longest diameter perpendicular to "A" (cm)].
4. Tumor burden must be completely encompassed by surgery or bleomycin-EPT.
5. Age: 18 years or older.
6. Men and women of childbearing potential must use physician approved contraceptive methods for 7 days following bleomycin-EPT.
7. Hematopoietic status:

   * Absolute neutrophil count (ANC) > 1000/uL
   * Platelets > 75,000/mm3
   * Prothrombin time:international normalized ratio (PT:INR) ? 1.5 (correctable with vitamin K injection)
8. Blood chemistry status:

   * Transaminases < 3 times upper limit of normal
   * Total bilirubin < 2.5 mg/dL
   * Creatinine < 2.5 mg/dL
9. A written Informed Consent form must be signed prior to the patient receiving any study procedures or treatments.

Exclusion Criteria:

1. Patients with tumors suspected of involving a 50% or greater encasement of a blood vessel as measured by magnetic resonance imaging (MRI) or computed tomography (CT) scan.
2. Patients with tumors having bone invasion.
3. Patients with any metallic implants in the treatment field.
4. Patients with hypersensitivity to bleomycin.
5. Patients who have received or will exceed a total lifetime dose of bleomycin greater than 400 units.
6. Patients deemed unsuitable for general anesthesia.
7. Patients with a significant history of emphysema or pulmonary fibrosis.
8. Patients with indwelling cardiac pacemakers who cannot tolerate a period with pacemaker turned off.
9. Patients with a history of uncontrolled cardiac arrhythmia.
10. Women who are pregnant, or are nursing. Women of childbearing potential must have a negative beta-human chorionic gonadotropin (beta-HCG) test within 7 days of study treatment.
11. Radiation therapy to the treatment area within 8 weeks of study treatment.
12. Chemotherapy or other cancer therapy (e.g., surgery, cryotherapy, etc.) to the treatment area within 4 weeks of study treatment.
13. Patients participating in a clinical study for an investigational drug or device within 4 weeks prior to the study treatment.
14. Patients previously randomized to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06-01 (Actual)

PRIMARY OUTCOMES:
Function status at 4 months using the performance status scale for head and neck cancer (PSSHN) and the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck (EORTC-QLC-H&N35) | 4 Months

SECONDARY OUTCOMES:
Local tumor recurrence, disease free survival and overall survival rates through 2 years after bleomycin-EPT or surgery treatment | 4 Months
Safety through 6 months after the study treatment | 6 Months
Durability of function status outcomes at 8 months after bleomycin-EPT or surgery treatment | 8 Months
Pharmacoeconomic parameters through 8 months after bleomycin-EPT or surgery treatment | 8 Months
Bleomycin systemic absorption and plasma pharmacokinetics following intratracheal (IT) bleomycin-EPT administration | 96 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goldfarb, MD, Study Chair — Inovio Pharmaceuticals
Locations (1):
- Inovio Biomedical Corporation, San Diego, California, United States